CLINICAL TRIAL: NCT01259479
Title: A Phase I Trial and Pharmacokinetic Study of the Oral Platinum Analog Satraplatin in Children and Young Adults With Refractory Solid Tumors Including Brain Tumors
Brief Title: Satraplatin in Children and Young Adults With Refractory Solid Tumors Including Brain Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 110047; 11-C-0047
Record Dates: First submitted 2010-12-11; First posted 2010-12-14 (Estimated); Last update posted 2018-07-05 (Actual); Status verified 2015-05-29

CONDITIONS: Solid Tumors; Brain Tumors; Brain Metastases
Keywords: Solid Tumors; Maximum Tolerated Dose; Parmacokinetics; Pharmacogenomics; Satraplatin; Cancer; Solid Tumor; Brain Tumor
MeSH Terms: conditions — Brain Neoplasms; Neoplasms | interventions — satraplatin

ARMS (1):
- 1 (Experimental): Dose escalation, continuous treatment without DLTs
  Interventions: Drug: Satraplatin

INTERVENTIONS:
Drug: Satraplatin — Orally, once daily for 5 days repeated every 28 days, dose-escalation

SUMMARY:
Background:

* Cisplatin and carboplatin are standard cancer treatment drugs used for various childhood cancers, including brain tumors. Both drugs frequently have severe side effects that may reduce their effectiveness, particularly in children, and new treatments are needed that may be similarly effective but less toxic for cancer patients.
* Satraplatin is an experimental drug, similar to cisplatin and carboplatin, that has not yet been approved by the Food and Drug Administration. Satraplatin has been shown to treat cancer by interfering with genetic material (DNA) in cancer cells. Some adults with cancer who have received satraplatin had slowing of the growth or shrinkage of their tumor. Researchers are interested in determining whether satraplatin can be effective for cancers that occur in children.

Objectives:

* To evaluate the safety and effectiveness of satraplatin as a treatment for children and young adults who have solid tumors that have not responded to standard treatment.
* To study the effects of satraplatin on the body in terms of side effects and blood chemistry.
* To examine the effect that genetic variations may have on the effectiveness of satraplatin.

Eligibility:

- Children, adolescents, and young adults between 3 and 21 years of age who have solid tumors (including brain tumors) that have not responded to standard treatment.

Design:

* Participants will be screened with a full physical examination and medical history, blood tests, and tumor imaging studies.
* Participants will receive satraplatin pills to be taken every day in the morning for 5 consecutive days, with no food for 2 hours before or 1 hour after the dose. Participants will then have 23 days without the drug to complete a 28-day cycle of treatment. Participants will also receive medication to prevent nausea and vomiting 30 minutes before the first dose of satraplatin. Following the first dose of satraplatin, medication for nausea will be given if needed.
* Satraplatin doses will be adjusted based on response to treatment, including potential side effects. Participants will have frequent blood tests and imaging studies to evaluate the effectiveness of the treatment and monitor any side effects, as well as hearing tests and other examinations as required by the study researchers.
* Participants will receive satraplatin every 4 weeks for up to 2 years until serious side effects occur or the tumor stops responding to treatment.

DETAILED DESCRIPTION:
BACKGROUND

The platinum compounds cisplatin and carboplatin are standard agents in the treatment of a variety of childhood cancers. However, cumulative and long-term renal and ototoxicity are a concern related to cisplatin administration, particularly in young children.

Several mechanisms of resistance to platinum compounds have been described including decreased drug accumulation due to altered drug uptake or the presence of a membrane efflux pump, increased intracellular levels of thiol-containing groups that detoxify and modulate platinum, and removal of the platinum-DNA adducts by DNA repair pathways called nucleotide excision repair (NER) and base excision repair (BER) pathways.

Polymorphisms in DNA repair genes have been shown in some cancers to predict better treatment response to platinum treatment.

Satraplatin is an oral platinum analog with similar preclinical in vitro and in vivo activity to that of cisplatin and carboplatin, and with activity in platinum resistant models.

Dose-limiting satraplatin toxicities in adults include nausea, vomiting, and myelosuppression. Neither renal nor neurologic toxicities have been described.

Satraplatin has demonstrated clinical activity in adult refractory tumors at the recommended phase II and III dose of 80 mg/m2/dose daily for 5 days every 28 or 35 days.

OBJECTIVES

To determine the maximum tolerated dose (MTD) of oral satraplatin administered on a once daily for 5 days every 28 days schedule in pediatric patients with relapsed or refractory solid tumors including brain tumors.

To define the toxicities of oral satraplatin and characterize the pharmacokinetics of oral satraplatin in children with refractory cancer.

To determine the preliminary antitumor activity of satraplatin.

To evaluate the pharmacogenomic expression of DNA repair genes in peripheral blood mononuclear blood cells.

ELIGIBILITY

Patients greater than or equal to 3 years and less than or equal to 25 years at enrollment with relapsed or refractory solid tumors including brain tumors.

Adequate organ function

DESIGN

This is a phase I trial of satraplatin administered once daily orally for 5 days every 28 days. A cycle of therapy is considered to be 28 days. The starting dose level is 60 mg/m(2)/dose with escalations to 80, 110, 140 mg/m(2)/dose. The MTD will be defined based on satraplatin tolerability during cycle one.

Disease status will be evaluated prior to every odd treatment cycle and therapy may continue for up to 2 years in the absence of progressive disease or unacceptable toxicity.

Plasma pharmacokinetics and pharmacogenomics will be evaluated during the first treatment cycle.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Age: greater than or equal to 3 years and less than or equal to 25 years of age at the time of study enrollment.
  2. Diagnosis: Patients with refractory solid tumors including brain tumors (including brain metastases). All patients must have had histological verification of the solid tumor at initial diagnosis or relapse with the exception of patients with diffuse intrinsic brainstem tumors, optic pathway tumors, or CNS germ cell tumors with elevations of reliable serum or CSF tumor markers (alpha-fetoprotein or beta-HCG).
  3. Disease status: Patients must have measurable or evaluable disease.
  4. Prior Therapy: Refractory to standard therapy and no other standard curative treatment options are available. Patients must have fully recovered to less than or equal to grade 1 from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering this study.

     i. Stem Cell Transplantation: Patients must be greater than or equal to 3 months since autologous stem cell transplant and greater than or equal to 6 months since allogeneic stem cell transplant prior to study entry.

     ii. Radiation Therapy: Extensive radiation therapy (craniospinal, more than half of the pelvis, TBI) must be completed at least 3 months prior to study entry. The last dose of all other local palliative radiation must be at least 2 weeks prior to study entry.

     iii. Myelosuppressive chemotherapy: The last dose of myelosuppressive chemotherapy must be at least 21 days prior to study entry. Therapy with nitrosoureas must be at least 6 weeks prior to study entry; and therapy with temozolomide must be 4 weeks prior to study entry.

     iv. Investigational anti-cancer agents: The last dose of all investigational agents must be at least 30 days prior to study entry.

     v. Growth factors: The last dose of growth factors such as filgrastim and epoetin must be at least one week prior to study entry. The last dose of long-acting colony stimulating factors, such as pegfilgrastim, must be 2 weeks prior to study entry.

     vi. Biologic anti-cancer agents: The last dose of nonmyelosuppressive biologic agents for the treatment of the patient s cancer must be at least 7 days prior to study entry.

     vii. Immunotherapy: At least 6 weeks since the completion of any type of immunotherapy, e.g. tumor vaccines.

     viii. Monoclonal antibody: At least 3 half-lives of the antibody after the last dose of a monoclonal antibody. (See table on Children s Oncology Group Phase I Consortium DVL homepage https://members.childrensoncologygroup.org/Disc/devtherapeu tics/default.asp for listing of monoclonal antibody half-lives.)

     ix. Corticosteroids: Patients with brain tumors must be on a stable or tapering dose of corticosteroids for 7 days prior to the date of the baseline scan performed for the purpose of assessing response to therapy on this study.
  5. Performance status: Patients greater than 10 years of age must have a Karnofsky performance level of greater than or equal to 50%, and children less than or equal to 10 years old must have a Lansky performance of greater than or equal to 50% (Appendix I). Patients who are wheelchair bound because of paralysis should be considered ambulatory when they are up in their wheel chair.
  6. Hematologic Function: Patients must have an absolute neutrophil count greater than or equal to 1000/microL, hemoglobin greater than or equal to 9g/dl (transfusion permitted), and platelet greater than or equal to 75,000/?l (transfusion independent).
  7. Hepatic Function: Patients must have bilirubin less than or equal to 1.5 times the upper limit of normal (ULN) for age, with the exception of Gilbert syndrome, and ALT within less than or equal to 3.0 times the ULN.
  8. Renal Function: Patients must have a creatinine clearance or radioisotope GFR greater than or equal to 60ml/min/1.73 m(2) or a normal serum creatinine based on age described below.
* Less than or equal to 5 years of age: a maximum serum creatinine of 0.8 mg/dL
* Older than 5 years of age but less than or equal to the age of 10: a maximum serum creatinine of 1.0 mg/dL
* Older than 10 years of age and less than or equal to the age of 15: a maximum serum creatinine of 1.2 mg/dL
* Older than 15 years of age: a maximum serum creatinine of 1.5 mg/dL

  9. Informed Consent: Diagnostic or laboratory studies performed exclusively to determine eligibility for this trial must only be done after obtaining written informed consent from all patients or their legal guardians (if the patient is <18 years old). When appropriate, pediatric patients will be included in all discussions. This can be accomplished through one of the following mechanisms:
  1. the NCI, POB screening protocol,
  2. an IRB-approved institutional screening protocol or
  3. the study-specific protocol.

     Documentation of the informed consent for screening will be maintained in the patient s research chart. Studies or procedures that were performed for clinical indications (not exclusively to determine eligibility) may be used for baseline values even if the studies were done before informed consent was obtained.

     10. Durable Power of Attorney (DPA): All patients >18 years of age will be offered the opportunity to assign DPA so that another person can make decisions about their medical care if they become incapacitated or cognitively impaired.

     EXCLUSION CRITERIA:
     1. Pregnant or breast-feeding females are excluded due to potential risks of fetal and teratogenic adverse events of an investigational agent. Pregnancy tests (urine BhCG) must be obtained prior to enrollment on this study in girls, age 9 years or older. Males or females of reproductive potential may not participate unless they have agreed to use an effective contraceptive method. Abstinence is an acceptable method of birth control.
     2. Last dose of any investigational agent given within the past 30 days. 3. Ongoing radiation therapy, chemotherapy, hormonal therapy directed at the tumor, immunotherapy, or biologic therapy.

     4. Active graft versus host disease.

     5. Graft vs Host Disease (GVHD) therapy or agents to prevent organ rejection post-transplant: Patients who are receiving cyclosporine, tacrolimus or other agents to prevent either GVHD post bone marrow transplant or organ rejection post transplant are not eligible for this trial.

     6. Clinically significant uncontrolled unrelated systemic illness such as serious infections or significant cardiac, pulmonary, hepatic or other organ dysfunction.

     7. Patients who in the opinion of the investigator may not be able to comply with the safety monitoring requirements of the study.

     8. Inability to swallow capsules as capsules cannot be crushed or broken

     9. Prior treatment with satraplatin.

Ages: 3 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 9 (Actual)
Dates: Start 2010-12-03; Primary Completion 2013-08-01 (Actual); Study Completion 2015-05-29 (Actual)

PRIMARY OUTCOMES:
MTD | 1 Year

SECONDARY OUTCOMES:
PKs | 1 Year
Definte anti-tumore activity | 1 Year
PGs | 1 Year

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte C Widemann, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Daw NC, Billups CA, Rodriguez-Galindo C, McCarville MB, Rao BN, Cain AM, Jenkins JJ, Neel MD, Meyer WH. Metastatic osteosarcoma. Cancer. 2006 Jan 15;106(2):403-12. doi: 10.1002/cncr.21626. PMID 16353204
- [Background] Ferguson WS, Harris MB, Goorin AM, Gebhardt MC, Link MP, Shochat SJ, Siegal GP, Devidas M, Grier HE. Presurgical window of carboplatin and surgery and multidrug chemotherapy for the treatment of newly diagnosed metastatic or unresectable osteosarcoma: Pediatric Oncology Group Trial. J Pediatr Hematol Oncol. 2001 Aug-Sep;23(6):340-8. doi: 10.1097/00043426-200108000-00004. PMID 11563767
- [Background] MacDonald TJ, Arenson EB, Ater J, Sposto R, Bevan HE, Bruner J, Deutsch M, Kurczynski E, Luerssen T, McGuire-Cullen P, O'Brien R, Shah N, Steinbok P, Strain J, Thomson J, Holmes E, Vezina G, Yates A, Phillips P, Packer R. Phase II study of high-dose chemotherapy before radiation in children with newly diagnosed high-grade astrocytoma: final analysis of Children's Cancer Group Study 9933. Cancer. 2005 Dec 15;104(12):2862-71. doi: 10.1002/cncr.21593. PMID 16315242